CLINICAL TRIAL: NCT06105879
Title: Can Transcutaneous Levels of Bilirubin Obtained From Covered Skin Replace Serum Bilirubin Measurement in Neonates Undergoing Phototherapy
Brief Title: Transcutaneous Bilirubin Levels From Covered Skin
Status: Completed | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Dilek Kahvecioğlu, Assoc. Prof., Ankara Training and Research Hospital
Other Study IDs: 1
Record Dates: First submitted 2023-10-12; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Hyperbilirubinemia, Neonatal
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: None Retained — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Serum: Total Serum bilirubin
  Interventions: Device: covered or open skin
- covered skin: Covered Skin Transcutaneous Bilirubin
  Interventions: Device: covered or open skin
- exposed skin: Exposed skin Transcutaneous Bilirubin
  Interventions: Device: covered or open skin

INTERVENTIONS:
Device: covered or open skin — transcutaneous mesarument of covered or open skin area

SUMMARY:
The aim of this study was to evaluate the levels of total serum bilirubin and transcutaneous bilirubin in newborns, measured in both covered and exposed areas, before phototherapy, 24th hour of phototherapy and 8 hours after cessation of phototherapy. The study included term and preterm newborns that required phototherapy between postnatal days 0-28. Total serum bilirubin levels and transcutaneous bilirubin measurements were obtained using the MBJ20-2019 Transcutaneous Handheld Bilirubinometer (Beijing M&B Electronic Instruments Co. Ltd. China, 2019) from both exposed (sternal) and unexposed (forehead, covered with a radio-opaque patch) areas before, at 24th hours and eight hours after phototherapy.

DETAILED DESCRIPTION:
Aim: This study aimed to evaluate total serum bilirubin and transcutaneous bilirubin levels measured from covered and exposed areas in newborns before phototherapy, after 24 hours of phototherapy, and 8 hours after discontinuing phototherapy.

Materials and Methods: Term and preterm newborns who needed phototherapy between postnatal days 0-28 were included in the study. Total serum bilirubin values and transcutaneous bilirubin measurements by MBJ20-2019 Transcutaneous Handheld Bilirubinometer (Beijing M&B Electronic Instruments Co. Ltd. China, 2019) from the exposed area (on sternum) and an unexposed area (forehead, covered with a radioopaque patch) were obtained before starting phototherapy, after 24 hours of phototherapy, and at 8 hours after phototherapy. The results were analyzed statistically using intraclass correlation coefficients (ICC).

ELIGIBILITY:
Inclusion Criteria:

Aged 0-28 days, Diagnosis of indirect hyperbilirubinemia Parent/guardian consent was obtained.

Exclusion Criteria:

Direct hyperbilirubinemia, Major congenital anomaly, Severe sepsis, Circulatory disorder, Need for blood exchange, Rehospitalization

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with indirect hyperbilirubinemia were admitted to the NICU
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
transcutaneous bilirubin levels measured from covered skin | first hour before phototherapy, after 24 hours of phototherapy, and 8 hours after discontinuing phototherapy.
  correlation between transcutaneous bilirubin levels measured from covered skin and total serum bilirubin measurements in newborns
transcutaneous bilirubin levels measured from open skin | first hour before phototherapy, after 24 hours of phototherapy, and 8 hours after discontinuing phototherapy.
  correlation between transcutaneous bilirubin levels measured from open skin and total serum bilirubin measurements in newborns

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Kahvecioglu, Assoc.Prof., Principal Investigator — Ankara Training and Research Hospital; Dilek Kahvecioglu, Assoc.Prof., Study Chair — Ankara Training and Research Hospital; Dilek Kahvecioglu, Assoc.Prof., Study Director — Ankara Training and Research Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided